CLINICAL TRIAL: NCT04610528
Title: A Window-of-opportunity Study of U3-1402, a HER3-targeting Antibody-drug Conjugate in Operable Breast Cancer According to ERBB3 Expression
Acronym: TOT-HER3
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SOLTI Breast Cancer Research Group (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOLTI-1805; 2019-004964-23 (EudraCT Number)
Record Dates: First submitted 2020-10-27; First posted 2020-10-30 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: HER3; antibody drug conjugate
MeSH Terms: conditions — Breast Neoplasms | interventions — patritumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- U3-1402 (Experimental): U3-1402 is an antibody drug conjugate (ADC) comprising a recombinant fully human anti-human epidermal growth factor receptor (HER) 3 immunoglobulin G1 (IgG1) monoclonal antibody (patritumab, U3-1287) covalently conjugated to a drug-linker (MAAA-1162a) containing a drug component (MAAA-1181a). MAAA-1181a is released after internalization and leads to apoptosis of the target tumor cells by the inhibition of topoisomerase I
  Interventions: Drug: U3 1402

INTERVENTIONS:
Drug: U3 1402 — 6.4 mg/kg dose
  Other Names: Patritumab Deruxtecan
Drug: U3 1402 — 5.6 mg/kg dose
  Other Names: Patritumab Deruxtecan

SUMMARY:
This is a prospective, multicenter, single arm, window-of-opportunity study evaluating the biological effect of U3-1402 in treatment naïve patients with early breast cancer, whose primary tumors are ≥1 cm by ultrasound evaluation.

The primary objective is to evaluate the biological activity of U3-1402, measured as the CelTIL score increase at post-treatment (C1D21) in HR+/HER2-negative BC included patients.

The study will consist of 2 parts enrolling ~115 patients.

* Part A will target to treat, with 6.4 mg/kg dose, 80 patients with HR-positive/HER2-negative tumors and
* Part B will target to treat with 5.6 mg/kg dose 20 patients with HR-positive/HER2-negative and 15 patients with TNBC tumors

Part A will test U3-1402 in patients with HR-positive/HER2-negative early breast cancer with a dose of 6.4 mg/kg. Part B will consist in testing 5.6 mg/kg dose of U3-1402 in patients with HR-positive/HER2-negative early breast cancer and in triple-negative early breast cancer and will be performed sequentially after Part A.

ELIGIBILITY:
Inclusion Criteria:

1. Written ICF for all study procedures according to local regulatory requirements prior to beginning specific protocol procedures.
2. Premenopausal or postmenopausal women and men, age ≥ 18 years.
3. ECOG Performance Status 0 - 1.
4. Histologically confirmed non-metastatic primary invasive adenocarcinoma of the breast untreated and recently diagnosed, with all the following characteristics:

   * At least one lesion that can be measured in at least 1 dimension with ≥ 1 cm in largest diameter measured by ultrasound.
   * Absence of distant metastasis (M0) as determined by institutional practice.
   * In the case of a multifocal tumor (defined as the presence of two or more foci of cancer within the same breast quadrant), the largest lesion must be ≥ 1 cm and designated the "target" lesion for all subsequent tumor evaluations and biopsies.
5. Patient must have biopsiable disease.
6. Only for HR+/HER2-negative patients: Estrogen (ER)-positive and/or Progesterone (PgR)-positive and HER2-negative tumor by the most recent American Society of Clinical Oncology - College of American Pathologists (ASCO-CAP) guidelines: ER and PgR defined as IHC nuclear staining ≥1% and HER2 negative locally assessed. Only for TNBC patients: Estrogen (ER)-negative and Progesterone (PgR)-negative and HER2-negative tumor by the most recent American Society of Clinical Oncology - College of American Pathologists (ASCO-CAP) guidelines: ER and PgR defined as IHC nuclear staining <1% and HER2 negative locally assessed
7. Ki67% ≥ 10% locally assessed (Dowsset et al. Journal of the National Cancer Institute, 103 (22), 1656-1664. 2011).
8. Available pre-treatment FFPE core needle biopsy evaluable for PAM50 and ERBB3 mRNA expression. Minimal sample requirements are to have at least 2 tumor cylinders with a minimal tissue surface of 10 mm2 tissue, containing at least 50% tumor cells and having enough tissue to do at least 20 cuts of 4 μm each. Macrodissection is allowed when needed. If archival tissue is either insufficient or unavailable, a new biopsy from the pretreated tumor must be obtained. Patients whose tumor tissue is not evaluable for ERBB3 expression central testing are not eligible.
9. Baseline LVEF ≥ 50% measured by echocardiography (ECHO) or Multiple Gate Acquisition (MUGA) scan
10. Adequate organ function, as determined by the following laboratory tests prior to randomization:

    * Hematological

      * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
      * Platelet count ≥ 100 x 109/L
      * Hemoglobin ≥ 9 g/dL (red blood cell transfusion and/or erythropoietin allowed)
    * Renal

      o Serum creatinine ≤ 1.5 x upper limit of normal (ULN), or 24-hour creatinine clearance ≥ 60 mL/min for subject with creatinine levels > 1.5 x ULN. (Note: Creatinine clearance does not need to be determined if the baseline serum creatinine is within normal limits. Creatinine clearance should be calculated per institutional standard).
    * Hepatic

      * Serum bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ ULN for a subject with total bilirubin level > 1.5 x ULN
      * Aspartate aminotransferase (AST) ≤ 3 x ULN
      * Alanine aminotransferase (ALT) ≤ 3 x ULN
      * Coagulation International normalization ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN
      * Partial thromboplastin time (PTT) or activated PTT (aPTT) ≤ 1.5 x ULN
11. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
12. Female subject of childbearing potential should have a negative urine or serum pregnancy test within 7 days prior to enrollment. If urine pregnancy test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Pregnancy testing does not need to be pursued in patients who are judged as postmenopausal before randomization, as determined by local practice, or who have undergone bilateral oophorectomy, total hysterectomy, or bilateral tubal ligation. Women of childbearing potential randomized to the treatment must use adequate contraception for the duration of protocol treatment and after 7 months after the study drug administration (see Appendix B).

Exclusion Criteria:

1. Inoperable locally advanced or inflammatory (i.e., inoperable Stage III) breast cancer.
2. Metastatic (Stage IV) breast cancer.
3. Bilateral invasive breast cancer.
4. Patients in whom a primary tumor excisional biopsy was performed.
5. Any prior treatment for primary actual invasive breast cancer.
6. Prior treatment with a HER3 antibody, topoisomerase I inhibitor, with an ADC which consists of an exatecan derivative that is a topoisomerase I inhibitor (e.g., DS-8201) and with a govitecan derivative (e.g., IMMU-132).
7. Medical history of symptomatic congestive heart failure (New York Heart Association classes II-IV) or serious cardiac arrhythmia requiring treatment; myocardial infarction within 6 months prior to randomization or unstable angina.
8. QT interval corrected using Fridericia's formula to > 450 millisecond (ms) in males and > 470 ms in females.
9. Any factors that increase the risk of corrected QT (QTc) interval prolongation or risk of arrhythmic events, such as congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives.
10. Medical history of clinically significant lung diseases (e.g., interstitial pneumonia, pneumonitis, pulmonary fibrosis, and severe radiation pneumonitis) or who are suspected to have these diseases by imaging at screening period.
11. Clinically significant corneal disease.
12. Major surgical procedure or significant traumatic injury within 28 days prior to randomization.
13. Assessment by the investigator to be unable or unwilling to comply with the requirements of the protocol.
14. History of other malignancy within the last 3 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other malignancies with an expected curative outcome.
15. Current severe, uncontrolled systemic disease (e.g. clinically significant cardiovascular, pulmonary or metabolic disease; wound healing disorders; ulcers; bone fractures).
16. Concurrent, serious, uncontrolled infections or current known infection with HIV or active hepatitis B and/or hepatitis C.
17. History of significant co-morbidities that, in the judgment of the investigator, may interfere with the conduction of the study, the evaluation of response, or with ICF.
18. Known hypersensitivity to either the drug substance components (including an antibody, a drug-linker, or a topoisomerase I inhibitor) or inactive ingredients in the drug product or history of severe hypersensitivity reactions to other monoclonal antibodies.
19. Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (i.e. pulmonary emboli within three months of the study enrollment, severe asthma, severe COPD, restrictive lung disease, pleural effusion etc.), and any autoimmune, connective tissue or inflammatory disorders with potential pulmonary involvement (i.e. rheumatoid arthritis, Sjögren's syndrome, sarcoidosis etc.), or prior pneumonectomy.
20. Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0, grade ≤1 or baseline. Subjects with chronic grade 2 toxicities may be eligible per the discretion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
CelTIL score | baseline and after one dose of U3-1402 at Cycle 1 Day 21
  Mean change in CelTIL score per central assessment in paired samples.
  CelTIL score = -0.8 × tumor cellularity (in %) + 1.3 × TILs (in %). The minimum and maximum unscaled CelTIL scores will be -80 and 130. This unscaled CelTIL score will then be scaled to reflect a range from 0 to 100 points.

SECONDARY OUTCOMES:
CelTIL score | baseline and after one dose of U3-1402 at Cycle 1 Day 21
  Mean change in CelTIL score per central assessment in paired samples for each ERBB3 cohort
ERBB3 levels vs. CelTIL score | baseline and after one dose of U3-1402 at Cycle 1 Day 21
  ERBB3 mRNA baseline levels and changes in CelTIL score for all patients and for each ERBB3 cohort
HER3 IHC vs. CelTIL score | baseline and after one dose of U3-1402 at Cycle 1 Day 21
  HER3 IHC baseline levels and changes in CelTIL score for all patients and for each ERBB3 cohort
PAM50 intrinsic subtypes vs. CelTIL score | baseline and after one dose of U3-1402 at Cycle 1 Day 21
  changes in CelTIL across the four PAM50 intrinsic subtypes.
Complete Cell Cycle Arrest (CCCA) | baseline and after one dose of U3-1402 at Cycle 1 Day 21
  determined per central assessment by IHC Ki67< 2.7%
ERBB3 mRNA expression vs. HER3 IHC | baseline
  Correlation coefficients between both biomarkers
safety and tolerability | through study completion, an average of 65 days each patient
  Type, incidence, severity (as graded by the NCI CTCAE v. 5.0), seriousness and attribution to the study medications of AEs and any laboratory abnormalities.
changes of HER3 expression. | t baseline, at Day 3-Day 7 (optional), Cycle 1 Day 21
  HER3 expression

CONTACTS AND LOCATIONS:
Locations (10):
- Spain (10):
  - ICO Badalona, Badalona, Barcelona
  - Institut Català d'Oncologia Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Centro Integral Oncológico Clara Campal (CIOCC), Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pascual T, Oliveira M, Ciruelos E, Bellet Ezquerra M, Saura C, Gavila J, Pernas S, Munoz M, Vidal MJ, Margeli Vila M, Cejalvo JM, Gonzalez-Farre B, Espinosa-Bravo M, Cruz J, Salvador-Bofill FJ, Guerra JA, Luna Barrera AM, Arumi de Dios M, Esker S, Fan PD, Martinez-Saez O, Villacampa G, Pare L, Ferrero-Cafiero JM, Villagrasa P, Prat A. SOLTI-1805 TOT-HER3 Study Concept: A Window-of-Opportunity Trial of Patritumab Deruxtecan, a HER3 Directed Antibody Drug Conjugate, in Patients With Early Breast Cancer. Front Oncol. 2021 Apr 23;11:638482. doi: 10.3389/fonc.2021.638482. eCollection 2021. PMID 33968735